CLINICAL TRIAL: NCT05540691
Title: Effect of Noise Blocking During General Anesthesia on Postoperative Pain in Patients Undergoing Laparoscopic Abdominal Surgery
Brief Title: Effect of Noise Blocking During General Anesthesia on Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Noise blocking and pain
Record Dates: First submitted 2022-09-06; First posted 2022-09-15 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2022-12

CONDITIONS: Postoperative Pain
Keywords: noise blocking; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients were randomly divided into intervention group（noise blocking） and control group（No noise blocking）
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): Intraoperative intervention with noise-canceling earphones was performed to isolate the noise
  Interventions: Device: Wear noise-cancelling earphones
- group 2 (No Intervention): After general anesthesia, the intervention of wearing noise-canceling earphones was not given

INTERVENTIONS:
Device: Wear noise-cancelling earphones — Intervention of wearing noise-canceling earphones after general anesthesia
  Arms: group 1

SUMMARY:
To investigate the effect of noise blocking during general anesthesia on postoperative pain in patients undergoing laparoscopic abdominal surgery. The aim of this study was to determine whether noise blocking can reduce postoperative pain, analgesic use, and its possible effects on intraoperative electrocorticogram.

ELIGIBILITY:
Inclusion Criteria:

* ASA Classification ⅰ-ⅲ
* Patients undergoing elective laparoscopic abdominal surgery under general anesthesia
* Voluntarily accept PCIA and signed informed consent

Exclusion Criteria:

* Patients with previous severe disease
* Patients with hearing abnormalities
* Patients requiring mechanical ventilation or undergoing epidural catheters or other types of regional anesthesia after surgery
* Patients with chronic preoperative pain and/or long-term analgesic use
* Patients who could not cooperate with the study for any reason

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-10-08 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Maximum pain score (NRS score) at 0-24 hours postoperatively | From ending of the surgery to 24 hours postoperatively
  NRS score: Pain was assessed on a scale of 0-10, with 0 being no pain and 10 being most painful
Pain score (NRS score) at 0-6 hours postoperatively | From ending of the surgery to 6 hours postoperatively
  NRS score: Pain was assessed on a scale of 0-10, with 0 being no pain and 10 being most painful
Pain score (NRS score) at 6-12 hours postoperatively | From 6 hours postoperatively to 12 hours postoperatively
  NRS score: Pain was assessed on a scale of 0-10, with 0 being no pain and 10 being most painful
Pain score (NRS score) at 12-24 hours postoperatively | From 12 hours postoperatively to 24 hours postoperatively
  NRS score: Pain was assessed on a scale of 0-10, with 0 being no pain and 10 being most painful

SECONDARY OUTCOMES:
Patient controlled analgesia pump analgesic consumption | From the time when the surgery was completed until to 24 hours after surgery
  Analgesic requirements was assessed by recording the volume of patient controlled analgesia pump
Postoperative hyperalgesia after surgery | from the 30 minutes before the surgery until to 30 minutes after surgery
  Postoperative hyperalgesia was measured by the ratio of pressure pain threshold at time when discharged from postanesthesia care unit compare to before surgery

CONTACTS AND LOCATIONS:
Overall Officials: Huang He, doctor, Study Chair — Department of Anesthesiology, The Second Affiliated Hospital, Chongqing Medical University
Locations (1):
- Department of Anesthesiology, The Second Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data for this study is available from the sponsor on reasonable request through email
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Five years after the study